CLINICAL TRIAL: NCT00390637
Title: Diet, Obesity and Genes
Brief Title: Diet, Obesity and Genes (DiOGenes)
Acronym: DIOGENES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Arne Astrup, Head of Department, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DiOGenes FP6-2005-513946; FOOD-2004-513946
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Metabolic Syndrome; Type 2 Diabetes; Cardiovascular Disease
Keywords: Diogenes; Diet Intervention; Family; Glycemic Index; Protein
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Low Protein, Low GI Diet
  Interventions: Behavioral: High or low Glycemic Index and high or low Protein Diet
- 2 (Experimental): Low Protein, High Glycemic Index Diet
  Interventions: Behavioral: High or low Glycemic Index and high or low Protein Diet
- 3 (Experimental): High Protein, Low Glycemic Index diet
  Interventions: Behavioral: High or low Glycemic Index and high or low Protein Diet
- 4 (Experimental): High Protein, High glycemic index diet
  Interventions: Behavioral: High or low Glycemic Index and high or low Protein Diet
- 5 (Experimental): Control diet (current recommendations)
  Interventions: Behavioral: High or low Glycemic Index and high or low Protein Diet

INTERVENTIONS:
Behavioral: High or low Glycemic Index and high or low Protein Diet

SUMMARY:
Study Title: Diogenes, A randomised controlled trial comparing the effect of reduced-fat diets varying in glycaemic index (high vs. low) and protein content (high vs. normal) on bodyweight in overweight and obese subjects after an initial weight loss.

DETAILED DESCRIPTION:
DiOGenes is a randomised controlled dietary intervention study in obese/overweight families (adults and children) in 8 different European countries, testing the efficacy and safety of diets differing in Glycaemic Index (GI) and protein content.

The 8 centres are divided into "shop centers" and "instruction centers", that provide different kind of dietary intervention and for a different length(see below):

The 2 Shop Centers (Denmark & The Netherlands):

Dietary periods and clinical examinations:

1. Clinical examination 1 with anthropometry, blood etc.
2. 8 week Low Calorie Diet (LCD) period (800-1000 kcal/day)(Adults only)
3. Clinical examination 2 with anthropometry, blood etc.
4. 6 months dietary intervention period 1 (SUPERMARKET period)(Family)
5. Clinical examination 3 with anthropometry, blood etc.
6. 6 months dietary intervention period 2 (DIETARY INSTRUCTION period)(Family).
7. Clinical examination 4 with anthropometry, blood ect.
8. 12 months free-living period with no dietary intervention. (Family)
9. Follow up (only body weight registration)

The 6 Instruction Centers (UK, Crete, Germany, Spain, Bulgaria, Czech Republic)

Dietary periods and clinical examinations:

1. Clinical examination 1 with anthropometry, blood etc.
2. 8 week Low Calorie Diet (LCD) period (800-1000 kcal/day). (Adults only)
3. Clinical examination 2 with anthropometry, blood etc.
4. 6 months dietary intervention period (DIETARY INSTRUCTION period). (Family)
5. Clinical examination 3 with anthropometry, blood etc.
6. 6 months free-living period with no dietary intervention. (Family)
7. Follow up (only body weight registration)

Note that, during the first 6 month intervention all families from the shop centers are provided all foods free of charge "SUPERMARKET PERIOD", whereas in the "Instruction Centers", the families receive dietary instruction only "Instruction Only".

ELIGIBILITY:
Inclusion Criteria:

* Families with healthy adults and children

Exclusion Criteria:

* Various

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
For adults: body weight loss maintenance | 6 Month
  The primary outcome is related to body weight loss maintenance after 6 month of intensive, homogeneous and therefore comparable dietary intervention across all 8 centres.

SECONDARY OUTCOMES:
For adults: change in body composition | 6 Month
  The relative loss or gain of fat mass and fat free mass
For adults: More than 5% weight loss maintenance | 6 month
  Achievement of 5% of body weight loss from randomization
For adults: More than 10% weight loss maintenance | 6 month
  Achievement of 10% of body weight loss from randomization
For adults: Drop out rate | 6 month
  Percentage drop out from randomisation to end of dietary intervention
For Adults: Change in risk factors for type-2 diabetes | 6 month
  Change in risk factors for type-2 diabetes
For Adults: Change in risk factors for cardiovascular disease | 6 month
  Change in risk factors for cardiovascular disease
For children: Change in body weight | 6 month
  Change in body weight from randomization to end of intervention
For Children: Change in BMI-Z-score | 6 month
  Change in BMI-Z-score from randomisation to end of intervention

OTHER OUTCOMES:
For adults: Identify traits biological that determine responses to the dietary intervention. | 12 months
  To identify biological traits that determine the family's and individual's responses to the dietary interventions.
For adults: Identify psychological traits that determine responses to the dietary intervention. | 12 months
  To identify psychological traits that determine the family's and individual's responses to the dietary interventions.
For adults: Identify traits gene - diet interactions that determine responses to the dietary intervention. | 12 months
  To identify gene - diet interactions (e.g. SNP x dietary intake or copy number x dietary intake) that determine the family's and individual's responses to the dietary interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Arne V Astrup, Professor, Principal Investigator — Institute of Human Nutrition, RVAU, Denmark
Locations (1):
- Arne V. Astrup, Copenhagen, Denmark

REFERENCES:
- [Background] Saris WH, Harper A. DiOGenes: a multidisciplinary offensive focused on the obesity epidemic. Obes Rev. 2005 May;6(2):175-6. doi: 10.1111/j.1467-789x.2005.00200.x. No abstract available. PMID 15836468
- [Derived] Grandjean P, Meddis A, Nielsen F, Astrup A, Budtz-Jorgensen E. Exposure to organochlorine compounds in relation to weight maintenance. Res Sq [Preprint]. 2025 Dec 12:rs.3.rs-8097114. doi: 10.21203/rs.3.rs-8097114/v1. PMID 41510295
- [Derived] Kemper EJ, Blaak EE, Adriaens ME, Meex RCR. Muscle and liver insulin resistance are associated with distinct plasma protein profiles; data from the DiOGenes trial. J Clin Endocrinol Metab. 2025 Oct 10:dgaf562. doi: 10.1210/clinem/dgaf562. Online ahead of print. PMID 41068881
- [Derived] Frances L, Croyal M, Ruidavets JB, Maraninchi M, Combes G, Raffin J, de Souto Barreto P, Ferrieres J, Blaak EE, Perret B, Moro C, Valero R, Martinez LO, Viguerie N. Identification of circulating apolipoprotein M as a new determinant of insulin sensitivity and relationship with adiponectin. Int J Obes (Lond). 2024 Jul;48(7):973-980. doi: 10.1038/s41366-024-01510-w. Epub 2024 Mar 15. PMID 38491190
- [Derived] Vidal-Ostos F, Ramos-Lopez O, Jebb SA, Papadaki A, Pfeiffer AFH, Handjieva-Darlenska T, Kunesova M, Blaak EE, Astrup A, Martinez JA; Diet, Obesity, and Genes (Diogenes) Project. Dietary protein and the glycemic index handle insulin resistance within a nutritional program for avoiding weight regain after energy-restricted induced weight loss. Nutr Metab (Lond). 2022 Oct 19;19(1):71. doi: 10.1186/s12986-022-00707-y. PMID 36261843
- [Derived] Imbert A, Vialaneix N, Marquis J, Vion J, Charpagne A, Metairon S, Laurens C, Moro C, Boulet N, Walter O, Lefebvre G, Hager J, Langin D, Saris WHM, Astrup A, Viguerie N, Valsesia A. Network Analyses Reveal Negative Link Between Changes in Adipose Tissue GDF15 and BMI During Dietary-induced Weight Loss. J Clin Endocrinol Metab. 2022 Jan 1;107(1):e130-e142. doi: 10.1210/clinem/dgab621. PMID 34415992
- [Derived] van der Kolk BW, Muniandy M, Kaminska D, Alvarez M, Ko A, Miao Z, Valsesia A, Langin D, Vaittinen M, Paakkonen M, Jokinen R, Kaye S, Heinonen S, Virtanen KA, Andersson DP, Mannisto V, Saris WH, Astrup A, Ryden M, Blaak EE, Pajukanta P, Pihlajamaki J, Pietilainen KH. Differential Mitochondrial Gene Expression in Adipose Tissue Following Weight Loss Induced by Diet or Bariatric Surgery. J Clin Endocrinol Metab. 2021 Apr 23;106(5):1312-1324. doi: 10.1210/clinem/dgab072. PMID 33560372
- [Derived] Ruffieux H, Carayol J, Popescu R, Harper ME, Dent R, Saris WHM, Astrup A, Hager J, Davison AC, Valsesia A. A fully joint Bayesian quantitative trait locus mapping of human protein abundance in plasma. PLoS Comput Biol. 2020 Jun 3;16(6):e1007882. doi: 10.1371/journal.pcbi.1007882. eCollection 2020 Jun. PMID 32492067
- [Derived] Turicchi J, O'Driscoll R, Finlayson G, Duarte C, Hopkins M, Martins N, Michalowska J, Larsen TM, van Baak MA, Astrup A, Stubbs RJ. Associations between the proportion of fat-free mass loss during weight loss, changes in appetite, and subsequent weight change: results from a randomized 2-stage dietary intervention trial. Am J Clin Nutr. 2020 Mar 1;111(3):536-544. doi: 10.1093/ajcn/nqz331. PMID 31950141
- [Derived] van der Kolk BW, Kalafati M, Adriaens M, van Greevenbroek MMJ, Vogelzangs N, Saris WHM, Astrup A, Valsesia A, Langin D, van der Kallen CJH, Eussen SJPM, Schalkwijk CG, Stehouwer CDA, Goossens GH, Arts ICW, Jocken JWE, Evelo CT, Blaak EE. Subcutaneous Adipose Tissue and Systemic Inflammation Are Associated With Peripheral but Not Hepatic Insulin Resistance in Humans. Diabetes. 2019 Dec;68(12):2247-2258. doi: 10.2337/db19-0560. Epub 2019 Sep 6. PMID 31492661
- [Derived] Valsesia A, Kulkarni SS, Marquis J, Leone P, Mironova P, Walter O, Hjorth MF, Descombes P, Hager J, Saris WH, Astrup A, Darimont C, O'Callaghan NJ. Salivary alpha-amylase copy number is not associated with weight trajectories and glycemic improvements following clinical weight loss: results from a 2-phase dietary intervention study. Am J Clin Nutr. 2019 Apr 1;109(4):1029-1037. doi: 10.1093/ajcn/nqy363. PMID 30982860
- [Derived] Svendstrup M, Allin KH, Angquist L, Schnohr P, Jensen GB, Linneberg A, Thuesen B, Astrup A, Saris WHM, Vestergaard H, Sorensen TIA. Is abdominal obesity at baseline influencing weight changes in observational studies and during weight loss interventions? Am J Clin Nutr. 2018 Nov 1;108(5):913-921. doi: 10.1093/ajcn/nqy187. PMID 30475965
- [Derived] Meyer A, Montastier E, Hager J, Saris WHM, Astrup A, Viguerie N, Valsesia A. Plasma metabolites and lipids predict insulin sensitivity improvement in obese, nondiabetic individuals after a 2-phase dietary intervention. Am J Clin Nutr. 2018 Jul 1;108(1):13-23. doi: 10.1093/ajcn/nqy087. PMID 29878058
- [Derived] Armenise C, Lefebvre G, Carayol J, Bonnel S, Bolton J, Di Cara A, Gheldof N, Descombes P, Langin D, Saris WH, Astrup A, Hager J, Viguerie N, Valsesia A. Transcriptome profiling from adipose tissue during a low-calorie diet reveals predictors of weight and glycemic outcomes in obese, nondiabetic subjects. Am J Clin Nutr. 2017 Sep;106(3):736-746. doi: 10.3945/ajcn.117.156216. Epub 2017 Aug 9. PMID 28793995
- [Derived] Hjorth MF, Ritz C, Blaak EE, Saris WH, Langin D, Poulsen SK, Larsen TM, Sorensen TI, Zohar Y, Astrup A. Pretreatment fasting plasma glucose and insulin modify dietary weight loss success: results from 3 randomized clinical trials. Am J Clin Nutr. 2017 Aug;106(2):499-505. doi: 10.3945/ajcn.117.155200. Epub 2017 Jul 5. PMID 28679551
- [Derived] Bolton J, Montastier E, Carayol J, Bonnel S, Mir L, Marques MA, Astrup A, Saris W, Iacovoni J, Villa-Vialaneix N, Valsesia A, Langin D, Viguerie N. Molecular Biomarkers for Weight Control in Obese Individuals Subjected to a Multiphase Dietary Intervention. J Clin Endocrinol Metab. 2017 Aug 1;102(8):2751-2761. doi: 10.1210/jc.2016-3997. PMID 28482007
- [Derived] Oller Moreno S, Cominetti O, Nunez Galindo A, Irincheeva I, Corthesy J, Astrup A, Saris WHM, Hager J, Kussmann M, Dayon L. The differential plasma proteome of obese and overweight individuals undergoing a nutritional weight loss and maintenance intervention. Proteomics Clin Appl. 2018 Jan;12(1). doi: 10.1002/prca.201600150. Epub 2017 May 15. PMID 28371297
- [Derived] Valsesia A, Saris WH, Astrup A, Hager J, Masoodi M. Distinct lipid profiles predict improved glycemic control in obese, nondiabetic patients after a low-caloric diet intervention: the Diet, Obesity and Genes randomized trial. Am J Clin Nutr. 2016 Sep;104(3):566-75. doi: 10.3945/ajcn.116.137646. Epub 2016 Aug 10. PMID 27510538
- [Derived] Navas-Carretero S, Holst C, Saris WH, van Baak MA, Jebb SA, Kafatos A, Papadaki A, Pfeiffer AF, Handjieva-Darlenska T, Hlavaty P, Stender S, Larsen TM, Astrup A, Martinez JA. The Impact of Gender and Protein Intake on the Success of Weight Maintenance and Associated Cardiovascular Risk Benefits, Independent of the Mode of Food Provision: The DiOGenes Randomized Trial. J Am Coll Nutr. 2016;35(1):20-30. doi: 10.1080/07315724.2014.948642. Epub 2015 Mar 31. PMID 25826291
- [Derived] Montastier E, Dejean S, Le Gall C, Saris WH, Langin D, Viguerie N. Adipose tissue CIDEA is associated, independently of weight variation, to change in insulin resistance during a longitudinal weight control dietary program in obese individuals. PLoS One. 2014 Jul 1;9(7):e98707. doi: 10.1371/journal.pone.0098707. eCollection 2014. PMID 24983748
- [Derived] Bendtsen LQ, Lorenzen JK, Larsen TM, van Baak M, Papadaki A, Martinez JA, Handjieva-Darlenska T, Jebb SA, Kunesova M, Pfeiffer AF, Saris WH, Astrup A, Raben A. Associations between dairy protein intake and body weight and risk markers of diabetes and CVD during weight maintenance. Br J Nutr. 2014 Mar 14;111(5):944-53. doi: 10.1017/S0007114513003322. Epub 2013 Oct 30. PMID 24168904
- [Derived] Damsgaard CT, Papadaki A, Jensen SM, Ritz C, Dalskov SM, Hlavaty P, Saris WH, Martinez JA, Handjieva-Darlenska T, Andersen MR, Stender S, Larsen TM, Astrup A, Molgaard C, Michaelsen KF; Diogenes. Higher protein diets consumed ad libitum improve cardiovascular risk markers in children of overweight parents from eight European countries. J Nutr. 2013 Jun;143(6):810-7. doi: 10.3945/jn.112.173427. Epub 2013 Apr 17. PMID 23596158
- [Derived] Papadaki A, Linardakis M, Plada M, Larsen TM, van Baak MA, Lindroos AK, Pfeiffer AF, Martinez JA, Handjieva-Darlenska T, Kunesova M, Holst C, Saris WH, Astrup A, Kafatos A; Diet, Obesity and Genes (DiOGenes) Project. A multicentre weight loss study using a low-calorie diet over 8 weeks: regional differences in efficacy across eight European cities. Swiss Med Wkly. 2013 Jan 21;143:w13721. doi: 10.4414/smw.2013.13721. eCollection 2013. PMID 23348658
- [Derived] Larsen LH, Angquist L, Vimaleswaran KS, Hager J, Viguerie N, Loos RJ, Handjieva-Darlenska T, Jebb SA, Kunesova M, Larsen TM, Martinez JA, Papadaki A, Pfeiffer AF, van Baak MA, Sorensen TIa, Holst C, Langin D, Astrup A, Saris WH. Analyses of single nucleotide polymorphisms in selected nutrient-sensitive genes in weight-regain prevention: the DIOGENES study. Am J Clin Nutr. 2012 May;95(5):1254-60. doi: 10.3945/ajcn.111.016543. Epub 2012 Apr 4. PMID 22492381
- [Derived] Gogebakan O, Kohl A, Osterhoff MA, van Baak MA, Jebb SA, Papadaki A, Martinez JA, Handjieva-Darlenska T, Hlavaty P, Weickert MO, Holst C, Saris WH, Astrup A, Pfeiffer AF; DiOGenes. Effects of weight loss and long-term weight maintenance with diets varying in protein and glycemic index on cardiovascular risk factors: the diet, obesity, and genes (DiOGenes) study: a randomized, controlled trial. Circulation. 2011 Dec 20;124(25):2829-38. doi: 10.1161/CIRCULATIONAHA.111.033274. Epub 2011 Nov 21. PMID 22104550
- [Derived] Mutch DM, Pers TH, Temanni MR, Pelloux V, Marquez-Quinones A, Holst C, Martinez JA, Babalis D, van Baak MA, Handjieva-Darlenska T, Walker CG, Astrup A, Saris WH, Langin D, Viguerie N, Zucker JD, Clement K; DiOGenes Project. A distinct adipose tissue gene expression response to caloric restriction predicts 6-mo weight maintenance in obese subjects. Am J Clin Nutr. 2011 Dec;94(6):1399-409. doi: 10.3945/ajcn.110.006858. Epub 2011 Oct 26. PMID 22030226
- [Derived] Rubio-Aliaga I, Marvin-Guy LF, Wang P, Wagniere S, Mansourian R, Fuerholz A, Saris WH, Astrup A, Mariman EC, Kussmann M. Mechanisms of weight maintenance under high- and low-protein, low-glycaemic index diets. Mol Nutr Food Res. 2011 Nov;55(11):1603-12. doi: 10.1002/mnfr.201100081. Epub 2011 Sep 29. PMID 21957032
- [Derived] Wang P, Holst C, Astrup A, Bouwman FG, van Otterdijk S, Wodzig WK, Andersen MR, van Baak MA, Rasmussen LG, Martinez JA, Jebb SA, Pfeiffer AF, Kafatos A, Handjieva-Darlenska T, Hlavaty P, Saris WH, Mariman EC; Diogenes Consortium. Blood profiling of proteins and steroids during weight maintenance with manipulation of dietary protein level and glycaemic index. Br J Nutr. 2012 Jan;107(1):106-19. doi: 10.1017/S0007114511002583. Epub 2011 Jun 23. PMID 21733334
- [Derived] Wang P, Holst C, Andersen MR, Astrup A, Bouwman FG, van Otterdijk S, Wodzig WK, van Baak MA, Larsen TM, Jebb SA, Kafatos A, Pfeiffer AF, Martinez JA, Handjieva-Darlenska T, Kunesova M, Saris WH, Mariman EC. Blood profile of proteins and steroid hormones predicts weight change after weight loss with interactions of dietary protein level and glycemic index. PLoS One. 2011 Feb 14;6(2):e16773. doi: 10.1371/journal.pone.0016773. PMID 21340022
- [Derived] Larsen TM, Dalskov SM, van Baak M, Jebb SA, Papadaki A, Pfeiffer AF, Martinez JA, Handjieva-Darlenska T, Kunesova M, Pihlsgard M, Stender S, Holst C, Saris WH, Astrup A; Diet, Obesity, and Genes (Diogenes) Project. Diets with high or low protein content and glycemic index for weight-loss maintenance. N Engl J Med. 2010 Nov 25;363(22):2102-13. doi: 10.1056/NEJMoa1007137. PMID 21105792
- [Derived] Papadaki A, Linardakis M, Larsen TM, van Baak MA, Lindroos AK, Pfeiffer AF, Martinez JA, Handjieva-Darlenska T, Kunesova M, Holst C, Astrup A, Saris WH, Kafatos A; DiOGenes Study Group. The effect of protein and glycemic index on children's body composition: the DiOGenes randomized study. Pediatrics. 2010 Nov;126(5):e1143-52. doi: 10.1542/peds.2009-3633. Epub 2010 Oct 11. PMID 20937657
- [Derived] Marquez-Quinones A, Mutch DM, Debard C, Wang P, Combes M, Roussel B, Holst C, Martinez JA, Handjieva-Darlenska T, Kalouskova P, Jebb S, Babalis D, Pfeiffer AF, Larsen TM, Astrup A, Saris WH, Mariman E, Clement K, Vidal H, Langin D, Viguerie N; DiOGenes Project. Adipose tissue transcriptome reflects variations between subjects with continued weight loss and subjects regaining weight 6 mo after caloric restriction independent of energy intake. Am J Clin Nutr. 2010 Oct;92(4):975-84. doi: 10.3945/ajcn.2010.29808. Epub 2010 Aug 25. PMID 20739421